CLINICAL TRIAL: NCT01076127
Title: Effect of Kettlebell Training on Musculoskeletal and Cardiovascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre for the Working Environment, Denmark (Other Government)
Responsible Party: Otto Melchior Poulsen, National Research Centre for the Working Environment, Denmark
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: VIMS02
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2010-12

CONDITIONS: Musculoskeletal Disorders
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketllebell group (Experimental): Basic ketllebell training 3 x 20 min a week for 8 weeks
  Interventions: Behavioral: Ketllebell training
- Control group (Sham Comparator): Control group. Receives a health examination before and after the intervention period, and are advised to stay active.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Ketllebell training — Kettlebell training 3 x 20 min a week for 8 weeks
  Arms: Ketllebell group
Behavioral: Control — Receives a health examination before and after the intervention period, and are advised to stay active.
  Arms: Control group

SUMMARY:
Neck/shoulder and back pain is quite common among employees in sedentary occupations. Furthermore, many have a low level of fitness. Strength training with dumbbells has been shown to alleviate neck/shoulder pain, but many people prefer to also have alternative training options. Empirically, kettlebell training works the neck/shoulder/back while at the same time training the cardiovascular system. This type of training has not previously been tested in a randomized controlled trial. The aim of this study is to test the effect of kettlebell training on musculoskeletal pain, fitness, and muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* employed
* office workers

Exclusion Criteria:

* trauma
* life threatening diseases
* pregnancy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Pain in the neck/shoulder and back | before and after the 8-week intervention
Muscle strength | before and after the 8-week intervention
Fitness (VO2-max) | before and after the 8-week intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lars L Andersen, PhD, Principal Investigator — National Research Centre for the Working Environment, Denmark
Locations (1):
- Novo Nordisk, Copenhagen, Denmark

REFERENCES:
- [Result] Jay K, Frisch D, Hansen K, Zebis MK, Andersen CH, Mortensen OS, Andersen LL. Kettlebell training for musculoskeletal and cardiovascular health: a randomized controlled trial. Scand J Work Environ Health. 2011 May;37(3):196-203. doi: 10.5271/sjweh.3136. Epub 2010 Nov 25. PMID 21107513
- See also: Our homepage — http://www.arbejdsmiljoforskning.dk